CLINICAL TRIAL: NCT03745469
Title: Effects of Smartphone Usage Duration on Neck Dysfunction in Young Versus Middle Aged Patients With Chronic Mechanical Neck Pain
Brief Title: The Effect of Smartphone Use Duration in Patients With Chronic Mechanical Neck Pain.
Status: Completed | Type: Observational
Sponsor: Aliaa Rehan Youssef (Other)
Responsible Party: Sponsor-Investigator, Aliaa Rehan Youssef, Associate Professor of Orthopedic Physical Therapy, Cairo University
Organization: Cairo University (Other)
Other Study IDs: Asmaa
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Neck Pain; Cervical Pain
Keywords: Smartphone; Age; proprioception; Deep cervical fatigue; neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young-age group: Patient between the age of 18 and 30 years old, with a confirmed diagnosis of chronic mechanical neck pain
  Interventions: Device: Smartphone
- Middle-age group: Patients between 30 and 60 years old, with a confirmed diagnosis of chronic mechanical neck pain.
  Interventions: Device: Smartphone

INTERVENTIONS:
Device: Smartphone — A standard smartphone will be used for browsing the internet for two different durations (10 and 30 minutes)
  Other Names: Smart phone; Cell phone; Mobile Phone

SUMMARY:
PURPOSE: The purpose of this study is to investigate the effects of smartphone usage duration on neck pain and sense of position as well as Deep Cervical Flexor (DCF) fatigue in young and middle aged patients with chronic mechanical neck pain.

BACKGROUND: Neck pain is one of most common causes of musculoskeletal disorders with a prevalence up to 86.8 %. It may interfere with the ability to perform normal activities of daily living (ADL). Patients with neck pain may present with reduced Rang of Motion (ROM) and diminished cervical position sense.

There are many risk factors that have been associated with neck pain including physiological factors such as age or pathomechanical factors such as increased physical demand on the spine. Smartphone use has been proposed as a risk factor for the development of neck pain in young adults due to sustaining a prolonged static posture or repeating particular neck movements for long period. The adverse effects of smartphone increases as the duration of the use increases. Aging is associated with increased cervical reposition error and reduced DCF muscle endurance, yet it is not clear how older adults will respond to prolonged use of smartphone.

HYPOTHESES: Increased duration of smartphone use will

1. increase neck pain in middle aged compared to young adult patients with chronic mechanical.
2. decrease cervical position sense in middle aged compared to young adult patients with chronic mechanical neck pain.
3. increase DCF fatigue in middle aged compared to young adult patients with chronic mechanical neck pain.

RESEARCH QUESTION: Would increased duration of smartphone usage accentuate neck pain, cervical reposition error and DCF fatigue in middle aged compared to young adults with chronic mechanical neck pain?

DETAILED DESCRIPTION:
Patients with chronic mechanical neck pain will be instructed to use a standard smartphone for web browsing, either for 10 or 30 minutes, while seated on a standard chair at two separate sessions. Task duration will be tested by a random order generated by the Excel software.

The outcome measures for this study will be neck pain, DCF fatigue and neck reposition error. All measures will be assessed prior to and immediately after performing the required task in each session by a single trained assessor.

Neck pain will be assessed using the visual analogue scale (VAS), proprioception acuity will be quantified by measuring the repositioning error angle using Cervical Range of Motion instrument (CROM) and DCF endurance will be quantified using the neck stabilizer pressure biofeedback device.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients with an age ranging from 18 to 60 years old.
2. Referred with a diagnosis of chronic mechanical neck pain for more than 3 months.
3. Patients should have at least a one year experience in using touch-screen smartphone.
4. Have a neck impairment of more than 8% on the neck disability index (NDI).

Exclusion Criteria:

1. Any history of upper extremity injury or surgery within the past year
2. Visual problems, dizziness and vertigo
3. Any deformity in the upper extremities or spine
4. Previous history of spinal surgery.
5. Neurological or systemic disorders that interfere with balance and sensation
6. Low back pain or deformity.
7. Patients with any red flags such as malignancy, infection, inflammation, myelopathy.
8. If patient having any physical difficulties interfering with the use of smartphone while sitting and standing.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity
Study Population: Patients will a confirmed diagnosis of chronic mechanical neck pain for over 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Current neck pain severity | 1 week
  Pain will be measured using the Visual Analogue Scale (VAS) which is a valid and reliable pain measurement tool.
  Each participant will be asked to put a mark on a 10-cm horizontal line that is marked with 'zero' at one end to indicate no pain and marked with'10' at the other end to indicate maximum pain.This ill be done at two separate session, before and immediately after using the smartphone for the specified period.

SECONDARY OUTCOMES:
DCF endurance | 1 week
  The endurance of DCF muscles will be assessed using the Neck stabilizer pressure biofeedback. This ill be done at two separate session, before and immediately after using the smartphone for the specified period.
Neck proprioception | 1 week
  repositioning error for neck flexion, extension and rotation will be measured using the CROM. Error will be calculated as absolute angle of error. This ill be done at two separate session, before and immediately after using the smartphone for the specified period.

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Rehan Youssef, PhD, Principal Investigator — Cairo University, Faculty of Physical Therapy
Locations (2):
- Egypt (2):
  - The outpatient clinic of the Faculty of Physical Therapy, Cairo University, Cairo
  - The outpatient Clinic, kasr Al-Aini Hospital, Cairo

IPD SHARING:
Plan to Share IPD: Undecided
Journal publications and conferences

REFERENCES:
- [Background] Adamo DE, Martin BJ, Brown SH. Age-related differences in upper limb proprioceptive acuity. Percept Mot Skills. 2007 Jun;104(3 Pt 2):1297-309. doi: 10.2466/pms.104.4.1297-1309. PMID 17879664
- [Background] AlAbdulwahab SS, Kachanathu SJ, AlMotairi MS. Smartphone use addiction can cause neck disability. Musculoskeletal Care. 2017 Mar;15(1):10-12. doi: 10.1002/msc.1170. Epub 2017 Jan 19. No abstract available. PMID 28105706
- [Background] Alahmari KA, Reddy RS, Silvian PS, Ahmad I, Kakaraparthi VN, Alam MM. Association of age on cervical joint position error. J Adv Res. 2017 May;8(3):201-207. doi: 10.1016/j.jare.2017.01.001. Epub 2017 Jan 9. PMID 28203459
- [Background] Almhdawi KA, Mathiowetz V, Al-Hourani Z, Khader Y, Kanaan SF, Alhasan M. Musculoskeletal pain symptoms among allied health professions' students: Prevalence rates and associated factors. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1291-1301. doi: 10.3233/BMR-169669. PMID 28946521
- [Background] AlZarea, B. K., & Patil, S. R. (2015). Mobile Phone Head and Neck Pain Syndrome : Proposal of a New Entity. Headache, 14(5), 63-3.
- [Background] Ariens GA, Bongers PM, Douwes M, Miedema MC, Hoogendoorn WE, van der Wal G, Bouter LM, van Mechelen W. Are neck flexion, neck rotation, and sitting at work risk factors for neck pain? Results of a prospective cohort study. Occup Environ Med. 2001 Mar;58(3):200-7. doi: 10.1136/oem.58.3.200. PMID 11171934
- [Background] Armstrong BS, McNair PJ, Williams M. Head and neck position sense in whiplash patients and healthy individuals and the effect of the cranio-cervical flexion action. Clin Biomech (Bristol). 2005 Aug;20(7):675-84. doi: 10.1016/j.clinbiomech.2005.03.009. PMID 15963617
- [Background] Arslan, Ahmet; Tutgun, A. (2013). Examination of cell phone usage habits and purposes of education faculty students. International Journal of Human Sciences, 10(1), 182-201.
- [Background] Audette I, Dumas JP, Cote JN, De Serres SJ. Validity and between-day reliability of the cervical range of motion (CROM) device. J Orthop Sports Phys Ther. 2010 May;40(5):318-23. doi: 10.2519/jospt.2010.3180. PMID 20436238
- [Background] Auffinger B, Lam S, Shen J, Thaci B, Roitberg BZ. Usefulness of minimum clinically important difference for assessing patients with subaxial degenerative cervical spine disease: statistical versus substantial clinical benefit. Acta Neurochir (Wien). 2013 Dec;155(12):2345-54; discussion 2355. doi: 10.1007/s00701-013-1909-4. Epub 2013 Oct 18. PMID 24136679
- [Background] Bababekova Y, Rosenfield M, Hue JE, Huang RR. Font size and viewing distance of handheld smart phones. Optom Vis Sci. 2011 Jul;88(7):795-7. doi: 10.1097/OPX.0b013e3182198792. PMID 21499163
- [Background] Binder A. The diagnosis and treatment of nonspecific neck pain and whiplash. Eura Medicophys. 2007 Mar;43(1):79-89. PMID 17369782
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Blatter, B. M., & Bongers, P. M. (2002). Duration of computer use and mouse use in relation to musculoskeletal disorders of neck or upper limb. International Journal of Industrial Ergonomics, 30(4-5), 295-306.
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932
- [Background] Boyd-Clark LC, Briggs CA, Galea MP. Muscle spindle distribution, morphology, and density in longus colli and multifidus muscles of the cervical spine. Spine (Phila Pa 1976). 2002 Apr 1;27(7):694-701. doi: 10.1097/00007632-200204010-00005. PMID 11923661
- [Background] Brink Y, Louw Q, Grimmer K, Jordaan E. The spinal posture of computing adolescents in a real-life setting. BMC Musculoskelet Disord. 2014 Jun 20;15:212. doi: 10.1186/1471-2474-15-212. PMID 24950887
- [Background] Cagnie B, Danneels L, Van Tiggelen D, De Loose V, Cambier D. Individual and work related risk factors for neck pain among office workers: a cross sectional study. Eur Spine J. 2007 May;16(5):679-86. doi: 10.1007/s00586-006-0269-7. Epub 2006 Dec 8. PMID 17160393
- [Background] Chiu TW, Lau KT, Ho CW, Ma MC, Yeung TF, Cheung PM. A study on the prevalence of and risk factors for neck pain in secondary school teachers. Public Health. 2006 Jun;120(6):563-5. doi: 10.1016/j.puhe.2006.01.007. Epub 2006 May 8. No abstract available. PMID 16684548
- [Background] Cleland JA, Fritz JM, Whitman JM, Palmer JA. The reliability and construct validity of the Neck Disability Index and patient specific functional scale in patients with cervical radiculopathy. Spine (Phila Pa 1976). 2006 Mar 1;31(5):598-602. doi: 10.1097/01.brs.0000201241.90914.22. PMID 16508559
- [Background] de Koning CH, van den Heuvel SP, Staal JB, Smits-Engelsman BC, Hendriks EJ. Clinimetric evaluation of active range of motion measures in patients with non-specific neck pain: a systematic review. Eur Spine J. 2008 Jul;17(7):905-21. doi: 10.1007/s00586-008-0656-3. Epub 2008 Apr 22. PMID 18427843
- [Background] Deschenes MR. Effects of aging on muscle fibre type and size. Sports Med. 2004;34(12):809-24. doi: 10.2165/00007256-200434120-00002. PMID 15462613
- [Background] Douglas, E. C., & Gallagher, K. M. (2018). Are the Neck Positions and Muscle Activity Observed when Reading a Tablet Similar to That of the Cervical Flexion-Relaxation Onset ? Are the Neck Positions and Muscle Activity Observed when Reading a Tablet Similar to That of the Cervical Flexion-Relaxati. IISE Transactions on Occupational Ergonomics and Human Factors, (Just-Accepted)., 1-7.
- [Background] Doumas M, Krampe RT. Adaptation and reintegration of proprioceptive information in young and older adults' postural control. J Neurophysiol. 2010 Oct;104(4):1969-77. doi: 10.1152/jn.00345.2010. Epub 2010 Aug 11. PMID 20702741
- [Background] Elwardany, S. H., El-sayed, W. H.,& Ali, M. F. . (2016). Validity of Kinovea Computer Program in Measuring Cervical Range of Motion in Frontal Plane, 84(1), 579-587.
- [Background] Xie YF, Szeto G, Madeleine P, Tsang S. Spinal kinematics during smartphone texting - A comparison between young adults with and without chronic neck-shoulder pain. Appl Ergon. 2018 Apr;68:160-168. doi: 10.1016/j.apergo.2017.10.018. Epub 2017 Nov 24. PMID 29409630
- [Background] Fletcher JP, Bandy WD. Intrarater reliability of CROM measurement of cervical spine active range of motion in persons with and without neck pain. J Orthop Sports Phys Ther. 2008 Oct;38(10):640-5. doi: 10.2519/jospt.2008.2680. PMID 18827326
- [Background] Florencio LL, Pereira PA, Silva ER, Pegoretti KS, Goncalves MC, Bevilaqua-Grossi D. Agreement and reliability of two non-invasive methods for assessing cervical range of motion among young adults. Rev Bras Fisioter. 2010 Mar-Apr;14(2):175-81. Epub 2010 May 14. English, Portuguese. PMID 20464161
- [Background] Gold JE, Driban JB, Thomas N, Chakravarty T, Channell V, Komaroff E. Postures, typing strategies, and gender differences in mobile device usage: an observational study. Appl Ergon. 2012 Mar;43(2):408-12. doi: 10.1016/j.apergo.2011.06.015. Epub 2011 Jul 20. PMID 21764031
- [Background] Gong, W., Kim, C., & Lee, Y. (2012). Correlations between Cervical Lordosis , Forward Head Posture , Cervical ROM and the Strength and Endurance of the Deep Neck Flexor Muscles in College Students. Journal of Physical Therapy Science, 24(3), 275-277.
- [Background] Goodpaster BH, Park SW, Harris TB, Kritchevsky SB, Nevitt M, Schwartz AV, Simonsick EM, Tylavsky FA, Visser M, Newman AB. The loss of skeletal muscle strength, mass, and quality in older adults: the health, aging and body composition study. J Gerontol A Biol Sci Med Sci. 2006 Oct;61(10):1059-64. doi: 10.1093/gerona/61.10.1059. PMID 17077199
- [Background] Green BN. A literature review of neck pain associated with computer use: public health implications. J Can Chiropr Assoc. 2008 Aug;52(3):161-7. PMID 18769599
- [Background] Greig, A. M., Straker, L. M., & Briggs, A. M. (2005). Cervical erector spinae and upper trapezius muscle activity in children using different information technologies. Physiotherapy, 91(2), 119-126.
- [Background] Guan X, Fan G, Chen Z, Zeng Y, Zhang H, Hu A, Gu G, Wu X, Gu X, He S. Gender difference in mobile phone use and the impact of digital device exposure on neck posture. Ergonomics. 2016 Nov;59(11):1453-1461. doi: 10.1080/00140139.2016.1147614. Epub 2016 Apr 5. PMID 27046745
- [Background] Guez M, Hildingsson C, Nilsson M, Toolanen G. The prevalence of neck pain: a population-based study from northern Sweden. Acta Orthop Scand. 2002 Aug;73(4):455-9. doi: 10.1080/00016470216329. PMID 12358121
- [Background] Hagberg M. ABC of work related disorders. Neck and arm disorders. BMJ. 1996 Aug 17;313(7054):419-22. doi: 10.1136/bmj.313.7054.419. No abstract available. PMID 8761237
- [Background] Harris KD, Heer DM, Roy TC, Santos DM, Whitman JM, Wainner RS. Reliability of a measurement of neck flexor muscle endurance. Phys Ther. 2005 Dec;85(12):1349-55. PMID 16305273
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Heikkila HV, Wenngren BI. Cervicocephalic kinesthetic sensibility, active range of cervical motion, and oculomotor function in patients with whiplash injury. Arch Phys Med Rehabil. 1998 Sep;79(9):1089-94. doi: 10.1016/s0003-9993(98)90176-9. PMID 9749689
- [Background] Hoy DG, Protani M, De R, Buchbinder R. The epidemiology of neck pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):783-92. doi: 10.1016/j.berh.2011.01.019. PMID 21665126
- [Background] Hudswell, S., Von Mengersen, M., & Lucas, N. (2005). The cranio-cervical flexion test using pressure biofeedback : A useful measure of cervical dysfunction in the clinical setting ? International Journal of Osteopathic Medicine, 8(3), 98-105.
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Hyong IH. The effects on dynamic balance of dual-tasking using smartphone functions. J Phys Ther Sci. 2015 Feb;27(2):527-9. doi: 10.1589/jpts.27.527. Epub 2015 Feb 17. PMID 25729208
- [Background] Izquierdo M, Hakkinen K, Anton A, Garrues M, Ibanez J, Ruesta M, Gorostiaga EM. Maximal strength and power, endurance performance, and serum hormones in middle-aged and elderly men. Med Sci Sports Exerc. 2001 Sep;33(9):1577-87. doi: 10.1097/00005768-200109000-00022. PMID 11528348
- [Background] Jerosch J, Prymka M. Proprioception and joint stability. Knee Surg Sports Traumatol Arthrosc. 1996;4(3):171-9. doi: 10.1007/BF01577413. PMID 8961235
- [Background] Johnston V, Jull G, Souvlis T, Jimmieson NL. Neck movement and muscle activity characteristics in female office workers with neck pain. Spine (Phila Pa 1976). 2008 Mar 1;33(5):555-63. doi: 10.1097/BRS.0b013e3181657d0d. PMID 18317202
- [Background] Johnston V, Jimmieson NL, Jull G, Souvlis T. Quantitative sensory measures distinguish office workers with varying levels of neck pain and disability. Pain. 2008 Jul 15;137(2):257-265. doi: 10.1016/j.pain.2007.08.037. Epub 2007 Oct 25. PMID 17964075
- [Background] Jull, G. A. (2000). Deep Cervical Flexor Muscle Dysfunction in Whiplash. Musculoskeletal Pain, 8(1-2), 143-154.
- [Background] Jun I, Kim K. A Comparison of the Deep Cervical Flexor Muscle Thicknesses in Subjects with and without Neck Pain during Craniocervical Flexion Exercises. J Phys Ther Sci. 2013 Nov;25(11):1373-5. doi: 10.1589/jpts.25.1373. Epub 2013 Dec 11. PMID 24396191
- [Background] Jung SI, Lee NK, Kang KW, Kim K, Lee DY. The effect of smartphone usage time on posture and respiratory function. J Phys Ther Sci. 2016 Jan;28(1):186-9. doi: 10.1589/jpts.28.186. Epub 2016 Jan 30. PMID 26957754
- [Background] Kalisch T, Kattenstroth JC, Kowalewski R, Tegenthoff M, Dinse HR. Age-related changes in the joint position sense of the human hand. Clin Interv Aging. 2012;7:499-507. doi: 10.2147/CIA.S37573. Epub 2012 Nov 22. PMID 23226011
- [Background] Kang JH, Park RY, Lee SJ, Kim JY, Yoon SR, Jung KI. The effect of the forward head posture on postural balance in long time computer based worker. Ann Rehabil Med. 2012 Feb;36(1):98-104. doi: 10.5535/arm.2012.36.1.98. Epub 2012 Feb 29. PMID 22506241
- [Background] Kietrys DM, Gerg MJ, Dropkin J, Gold JE. Mobile input device type, texting style and screen size influence upper extremity and trapezius muscle activity, and cervical posture while texting. Appl Ergon. 2015 Sep;50:98-104. doi: 10.1016/j.apergo.2015.03.003. Epub 2015 Mar 25. PMID 25959323
- [Background] Kim HJ; DH; Kim JS. The relationship between smartphone use and subjective musculoskeletal symptoms and university students. J Phys Ther Sci. 2015 Mar;27(3):575-9. doi: 10.1589/jpts.27.575. Epub 2015 Mar 31. PMID 25931684
- [Background] Kim JY, Kwag KI. Clinical effects of deep cervical flexor muscle activation in patients with chronic neck pain. J Phys Ther Sci. 2016 Jan;28(1):269-73. doi: 10.1589/jpts.28.269. Epub 2016 Jan 30. PMID 26957772
- [Background] Kim MS. Influence of neck pain on cervical movement in the sagittal plane during smartphone use. J Phys Ther Sci. 2015 Jan;27(1):15-7. doi: 10.1589/jpts.27.15. Epub 2015 Jan 9. PMID 25642027
- [Background] Ko, Kyung, Hee-Soo Kim, and J.-H. W. (2013). The Study of Muscle Fatigue and Risks of Musculoskeletal System Disorders from Text Inputting on a Smartphone. The Ergonomics Society of Korea, 32(3), 273-278.
- [Background] Ko PH, Hwang YH, Liang HW. Influence of smartphone use styles on typing performance and biomechanical exposure. Ergonomics. 2016 Jun;59(6):821-8. doi: 10.1080/00140139.2015.1088075. Epub 2015 Nov 3. PMID 26328936
- [Background] Kuo YL, Tully EA, Galea MP. Video analysis of sagittal spinal posture in healthy young and older adults. J Manipulative Physiol Ther. 2009 Mar-Apr;32(3):210-5. doi: 10.1016/j.jmpt.2009.02.002. PMID 19362231
- [Background] Kwon M, Kim DJ, Cho H, Yang S. The smartphone addiction scale: development and validation of a short version for adolescents. PLoS One. 2013 Dec 31;8(12):e83558. doi: 10.1371/journal.pone.0083558. eCollection 2013. PMID 24391787
- [Background] Kwon M, Lee JY, Won WY, Park JW, Min JA, Hahn C, Gu X, Choi JH, Kim DJ. Development and validation of a smartphone addiction scale (SAS). PLoS One. 2013;8(2):e56936. doi: 10.1371/journal.pone.0056936. Epub 2013 Feb 27. PMID 23468893
- [Background] Larsson B, Sogaard K, Rosendal L. Work related neck-shoulder pain: a review on magnitude, risk factors, biochemical characteristics, clinical picture and preventive interventions. Best Pract Res Clin Rheumatol. 2007 Jun;21(3):447-63. doi: 10.1016/j.berh.2007.02.015. PMID 17602993
- [Background] Lee H, Nicholson LL, Adams RD. Neck muscle endurance, self-report, and range of motion data from subjects with treated and untreated neck pain. J Manipulative Physiol Ther. 2005 Jan;28(1):25-32. doi: 10.1016/j.jmpt.2004.12.005. PMID 15726032
- [Background] Lee J, Seo K. The comparison of cervical repositioning errors according to smartphone addiction grades. J Phys Ther Sci. 2014 Apr;26(4):595-8. doi: 10.1589/jpts.26.595. Epub 2014 Apr 23. PMID 24764641
- [Background] Lee KA, Kieckhefer GM. Measuring human responses using visual analogue scales. West J Nurs Res. 1989 Feb;11(1):128-32. doi: 10.1177/019394598901100111. No abstract available. PMID 2728416
- [Background] Lee S, Kang H, Shin G. Head flexion angle while using a smartphone. Ergonomics. 2015;58(2):220-6. doi: 10.1080/00140139.2014.967311. Epub 2014 Oct 17. PMID 25323467
- [Background] Lee, S. Y., Lee, D. H., & Han, S. K. (2016). The Effects of Posture on Neck Flexion Angle While Using a Smartphone according to Duration. Korean Society of Physical Medicine, 11(3), 35-39.
- [Background] Lee TH, Liu TY. Postural and muscular responses while viewing different heights of screen. Int J Occup Saf Ergon. 2013;19(2):251-8. doi: 10.1080/10803548.2013.11076982. PMID 23759195
- [Background] Lee, C., & Lee, S. J. (2017). Prevalence and predictors of smartphone addiction proneness among Korean adolescents. Children and Youth Services Review, 77(4), 10-17.
- [Background] Lee, H. (2016). Neck Pain and Functioning in Daily Activities Associated with Smartphone Usage. Journal of Korean Physical Therapy, 28(3), 183-188.
- [Background] Lee HY, Wang JD, Yao G, Wang SF. Association between cervicocephalic kinesthetic sensibility and frequency of subclinical neck pain. Man Ther. 2008 Oct;13(5):419-25. doi: 10.1016/j.math.2007.04.001. Epub 2007 Jun 4. PMID 17544825
- [Background] Lee, S., Lee, P. T. D., & Han, P. T. S. (2016). The Effects of Posture on Neck Flexion Angle While Using a Smartphone according to Duration, 11(3), 35-39.
- [Background] Lin IM, Peper E. Psychophysiological patterns during cell phone text messaging: a preliminary study. Appl Psychophysiol Biofeedback. 2009 Mar;34(1):53-7. doi: 10.1007/s10484-009-9078-1. Epub 2009 Feb 6. PMID 19199025
- [Background] Loudon JK, Ruhl M, Field E. Ability to reproduce head position after whiplash injury. Spine (Phila Pa 1976). 1997 Apr 15;22(8):865-8. doi: 10.1097/00007632-199704150-00008. PMID 9127919
- [Background] Maroufi N, Ahmadi A, Mousavi Khatir SR. A comparative investigation of flexion relaxation phenomenon in healthy and chronic neck pain subjects. Eur Spine J. 2013 Jan;22(1):162-8. doi: 10.1007/s00586-012-2517-3. Epub 2012 Oct 1. PMID 23053754
- [Background] Nagai T, Abt JP, Sell TC, Clark NC, Smalley BW, Wirt MD, Lephart SM. Neck proprioception, strength, flexibility, and posture in pilots with and without neck pain history. Aviat Space Environ Med. 2014 May;85(5):529-35. doi: 10.3357/asem.3874.2014. PMID 24834567
- [Background] Narici MV, Maganaris CN, Reeves ND, Capodaglio P. Effect of aging on human muscle architecture. J Appl Physiol (1985). 2003 Dec;95(6):2229-34. doi: 10.1152/japplphysiol.00433.2003. Epub 2003 Jul 3. PMID 12844499
- [Background] Neupane, S., Ali, U. T. I., Mathew, A., & College, M. V. S. (2017). Text Neck Syndrome - Systematic Review. Imperial Journal of Interdisciplinary Research, 3(7), 141-148.
- [Background] O'Leary S, Falla D, Jull G. The relationship between superficial muscle activity during the cranio-cervical flexion test and clinical features in patients with chronic neck pain. Man Ther. 2011 Oct;16(5):452-5. doi: 10.1016/j.math.2011.02.008. Epub 2011 Mar 10. PMID 21396876
- [Background] Olaogun, M. O., Adedoyin, R. A., Ikem, I. C., & Anifaloba, O. R. (2004). Reliability of rating low back pain with a visual analogue scale and a semantic differential scale. Physiotherapy Theory and Practice, 20(2), 135-142.
- [Background] Lee S, Lee D, Park J. Effect of the cervical flexion angle during smart phone use on muscle fatigue of the cervical erector spinae and upper trapezius. J Phys Ther Sci. 2015 Jun;27(6):1847-9. doi: 10.1589/jpts.27.1847. Epub 2015 Jun 30. PMID 26180333
- [Background] Park, J., Kim, K., Kim, N., Choi, I., & Lee, S. (2015). A Comparison of Cervical Flexion , Pain , and Clinical Depression in Frequency of Smartphone Use. International Journal of Bio-Science and Bio-Technology, 7(3), 183-190.
- [Background] Park YH, An CM, Moon SJ. Effects of visual fatigue caused by smartphones on balance function in healthy adults. J Phys Ther Sci. 2017 Feb;29(2):221-223. doi: 10.1589/jpts.29.221. Epub 2017 Feb 24. PMID 28265143
- [Background] Patten CJ, Kircher A, Ostlund J, Nilsson L. Using mobile telephones: cognitive workload and attention resource allocation. Accid Anal Prev. 2004 May;36(3):341-50. doi: 10.1016/S0001-4575(03)00014-9. PMID 15003578
- [Background] Paul-Dauphin A, Guillemin F, Virion JM, Briancon S. Bias and precision in visual analogue scales: a randomized controlled trial. Am J Epidemiol. 1999 Nov 15;150(10):1117-27. doi: 10.1093/oxfordjournals.aje.a009937. PMID 10568628
- [Background] Peper, E., Waderich, K., Harvey, R., & Sutter, S. (2013). The Psychophysiology of Contemporary Information Technologies Tablets and Smartphones Can Be a Pain in the Neck 1. In Applied Psychophysiology and Biofeedback, 38(3), 219-233.
- [Background] Petersen, C. M., Zimmermann, C. L., & Tang, R. (2013). Proprioception interventions to improve cervical position sense in cervical pathology. International Journal of Therapy and Rehabilitation, 20(3), 154-163.
- [Background] Portelli A, Reid SA. Cervical Proprioception in a Young Population Who Spend Long Periods on Mobile Devices: A 2-Group Comparative Observational Study. J Manipulative Physiol Ther. 2018 Feb;41(2):123-128. doi: 10.1016/j.jmpt.2017.10.004. Epub 2018 Jan 17. PMID 29338884
- [Background] Rafat, D., Azab, E., Amin, D. I., Mohamed, G. I., Rafat, D., & Azab, E. (2017). Effect of smart phone using duration and gender on dynamic balance. International Journal of Medical Research & Health Sciences, 6(1), 42-49.
- [Background] Reddy, R. S., Maiya, G. A., & Rao, S. K. (2012). Proprioceptive reposition errors in subjects with cervical spondylosis. International Journal of Health Sciences & Research, 1(2), 65-73.
- [Background] Rix GD, Bagust J. Cervicocephalic kinesthetic sensibility in patients with chronic, nontraumatic cervical spine pain. Arch Phys Med Rehabil. 2001 Jul;82(7):911-9. doi: 10.1053/apmr.2001.23300. PMID 11441377
- [Background] Robbins S, Waked E, McClaran J. Proprioception and stability: foot position awareness as a function of age and footwear. Age Ageing. 1995 Jan;24(1):67-72. doi: 10.1093/ageing/24.1.67. PMID 7762465
- [Background] Ruivo RM, Pezarat-Correia P, Carita AI. Cervical and shoulder postural assessment of adolescents between 15 and 17 years old and association with upper quadrant pain. Braz J Phys Ther. 2014 Jul-Aug;18(4):364-71. doi: 10.1590/bjpt-rbf.2014.0027. Epub 2014 Jul 18. PMID 25054381
- [Background] Shaheen AA, Omar MT, Vernon H. Cross-cultural adaptation, reliability, and validity of the Arabic version of neck disability index in patients with neck pain. Spine (Phila Pa 1976). 2013 May 1;38(10):E609-15. doi: 10.1097/BRS.0b013e31828b2d09. PMID 23429690
- [Background] Shin H, Kim K. Effects of Cervical Flexion on the Flexion-relaxation Ratio during Smartphone Use. J Phys Ther Sci. 2014 Dec;26(12):1899-901. doi: 10.1589/jpts.26.1899. Epub 2014 Dec 25. PMID 25540493
- [Background] Silva AG, Punt TD, Sharples P, Vilas-Boas JP, Johnson MI. Head posture and neck pain of chronic nontraumatic origin: a comparison between patients and pain-free persons. Arch Phys Med Rehabil. 2009 Apr;90(4):669-74. doi: 10.1016/j.apmr.2008.10.018. PMID 19345785
- [Background] Sokka T. Assessment of pain in rheumatic diseases. Clin Exp Rheumatol. 2005 Sep-Oct;23(5 Suppl 39):S77-84. PMID 16273789
- [Background] Stanton TR, Leake HB, Chalmers KJ, Moseley GL. Evidence of Impaired Proprioception in Chronic, Idiopathic Neck Pain: Systematic Review and Meta-Analysis. Phys Ther. 2016 Jun;96(6):876-87. doi: 10.2522/ptj.20150241. Epub 2015 Oct 15. PMID 26472296
- [Background] Sterling M, Jull G, Wright A. The effect of musculoskeletal pain on motor activity and control. J Pain. 2001 Jun;2(3):135-45. doi: 10.1054/jpai.2001.19951. PMID 14622823
- [Background] Szeto, G. P. Y., Straker, L. M., & O'Sullivan, P. B. (2005). The effects of speed and force of keyboard operation on neck-shoulder muscle activities in symptomatic and asymptomatic office workers. International Journal of Industrial Ergonomics, 35(5), 429-444.